CLINICAL TRIAL: NCT01226927
Title: The Efficacy of Automated Intermittent Boluses for Continuous Femoral Nerve Block: a Prospective, Randomized Comparison to Continuous Infusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Larry C. Field, M.D., Department of Anesthesia and Perioperative Medicine, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR 18880
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Arthroplasty, Replacement, Knee; Nerve Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous infusion rate (Active Comparator): Patients received a continuous infusion of 0.2% ropivacaine at 10.1 mL/hr via their femoral nerve catheter.
  Interventions: Other: Automated intermittent bolus

INTERVENTIONS:
Other: Automated intermittent bolus — Automated intermittent bolus delivery method of 0.2% ropivacaine at 5 mL every 30 minutes with a basal infusion of 0.1 mL/hr.

SUMMARY:
The optimal infusion technique (continuous rate vs. intermittent bolus) for peripheral nerve blocks has not been established. To our knowledge, this is the first study to compare the efficacy of an automated intermittent bolus technique to a continuous rate of infusion of local anesthetic in femoral nerve catheters. We hypothesized that the intermittent bolus technique would provide enhanced analgesia compared to a continuous infusion rate as assessed by intravenous patient-controlled analgesia (IV-PCA) hydromorphone consumption and visual analog scale (VAS) pain scores.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1 through 3
* elective, primary, unilateral TKA

Exclusion Criteria:

* patient refusal
* pregnancy
* diabetic neuropathy or any other neurologic or neuromuscular disease
* rheumatoid arthritis
* current coagulopathy
* skin infection at needle insertion site for the femoral or sciatic blocks
* significant renal or hepatic impairment
* unsuccessful femoral or sciatic block or femoral catheter placement
* femoral catheter dislodgement after placement
* inability to understand VAS pain scales
* inability to use an IV-PCA pump

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Intravenous patient-controlled analgesia opioid consumption | Cumulative IV-PCA use was recorded until femoral nerve catheter removed on postoperative day 2.
Visual analog pain scale score | Preop; Immediately postoperatively in PACU; Postoperative day (POD) 0 at 8pm; POD 1 at 8am, 2pm & 8pm; POD 2 at 8am

SECONDARY OUTCOMES:
Visual analog scale patient satisfaction scores | POD 1 at 8am; POD 2 at 8am
Incidence of physician administered "rescue" boluses of the femoral nerve catheter
Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Larry C. Field, M.D., Principal Investigator — Department of Anesthesia and Perioperative Medicine, Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Chelly JE, Greger J, Gebhard R, Coupe K, Clyburn TA, Buckle R, Criswell A. Continuous femoral blocks improve recovery and outcome of patients undergoing total knee arthroplasty. J Arthroplasty. 2001 Jun;16(4):436-45. doi: 10.1054/arth.2001.23622. PMID 11402405
- [Background] Shum CF, Lo NN, Yeo SJ, Yang KY, Chong HC, Yeo SN. Continuous femoral nerve block in total knee arthroplasty: immediate and two-year outcomes. J Arthroplasty. 2009 Feb;24(2):204-9. doi: 10.1016/j.arth.2007.09.014. Epub 2008 Mar 4. PMID 18534496
- [Background] Lim Y, Sia AT, Ocampo C. Automated regular boluses for epidural analgesia: a comparison with continuous infusion. Int J Obstet Anesth. 2005 Oct;14(4):305-9. doi: 10.1016/j.ijoa.2005.05.004. PMID 16154735
- [Background] Wong CA, Ratliff JT, Sullivan JT, Scavone BM, Toledo P, McCarthy RJ. A randomized comparison of programmed intermittent epidural bolus with continuous epidural infusion for labor analgesia. Anesth Analg. 2006 Mar;102(3):904-9. doi: 10.1213/01.ane.0000197778.57615.1a. PMID 16492849
- [Background] Taboada M, Rodriguez J, Bermudez M, Amor M, Ulloa B, Aneiros F, Sebate S, Cortes J, Alvarez J, Atanassoff PG. Comparison of continuous infusion versus automated bolus for postoperative patient-controlled analgesia with popliteal sciatic nerve catheters. Anesthesiology. 2009 Jan;110(1):150-4. doi: 10.1097/ALN.0b013e318191693a. PMID 19104182
- [Background] Ferrante FM, Orav EJ, Rocco AG, Gallo J. A statistical model for pain in patient-controlled analgesia and conventional intramuscular opioid regimens. Anesth Analg. 1988 May;67(5):457-61. PMID 3364765
- [Background] Taboada M, Rodriguez J, Bermudez M, Valino C, Ulloa B, Aneiros F, Gude F, Cortes J, Alvarez J, Atanassoff PG. A "new" automated bolus technique for continuous popliteal block: a prospective, randomized comparison with a continuous infusion technique. Anesth Analg. 2008 Oct;107(4):1433-7. doi: 10.1213/ane.0b013e3181824164. PMID 18806065
- [Derived] Hillegass MG, Field LC, Stewart SR, Borckardt JJ, Dong L, Kotlowski PE, Demos HA, Del Schutte H, Reeves ST. The efficacy of automated intermittent boluses for continuous femoral nerve block: a prospective, randomized comparison to continuous infusions. J Clin Anesth. 2013 Jun;25(4):281-8. doi: 10.1016/j.jclinane.2012.11.015. Epub 2013 May 16. PMID 23685099